CLINICAL TRIAL: NCT04634864
Title: tDCS in Post-stroke Fatigue: a Double Blind, Sham-controlled, Bilateral Anodal Motor Cortical Stimulation Study
Brief Title: Transcranial Direct Current Stimulation in Post-stroke Fatigue
Acronym: TIPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 195246
Record Dates: First submitted 2020-11-12; First posted 2020-11-18 (Actual); Last update posted 2020-11-18 (Actual); Status verified 2020-11

CONDITIONS: Fatigue; Stroke
MeSH Terms: conditions — Fatigue; Stroke | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Anodal tDCS (Active Comparator): 40 minutes of 2mA intensity direct current stimulation
  Interventions: Device: Anodal tDCS
- sham tDCS (Sham Comparator): 40 minutes of 0mA intensity. the session starts with a ramp up to 2mA, but machine is switched off after 2 minutes of stimulation.
  Interventions: Device: sham tDCS

INTERVENTIONS:
Device: Anodal tDCS — 40 minutes of 2mA intensity direct current stimulation was delivered over both the right and left motor cortex simultaneously
  Arms: Anodal tDCS
Device: sham tDCS — The stimulator was switched off after 2 minutes of stimulation.
  Arms: sham tDCS

SUMMARY:
This is a double-blind, sham-controlled, anodal tDCS study to understand the effect of increasing motor cortex excitability on post-stroke fatigue.

ELIGIBILITY:
Inclusion Criteria:

Diagnosed with stroke at least 3 months post-stroke

Exclusion Criteria:

Other neurological conditions on Anti-depressants severe motor impairment (affected hand grip <60% unaffected hand) severe cognitive impairment (unable to follow instructions, or give informed consent) scored >11 in the depression sub-section of HADS questionnaire contraindications for TMS or tES

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2018-01-10 (Actual); Primary Completion 2019-08-08 (Actual); Study Completion 2019-08-08 (Actual)

PRIMARY OUTCOMES:
Fatigue Severity Scale - 7 | 2 weeks
  a questionnaire based fatigue scale

SECONDARY OUTCOMES:
Resting Motor Threshold | 1 day
  This is a measure of cortical excitability as measured by transcranial magnetic stimulation
Input-output curves | 1 day
  This is a measure of cortical recruitment as measured by transcranial magnetic stimulation
Perceived effort - Explicit | 1 day
  A VAS scale associated with a grip task
Perceived effort - Implicit | 1 day
  A novel line length estimation task

CONTACTS AND LOCATIONS:
Locations (1):
- 33 Queen Square, Institute of Neurology, UCL, London, United Kingdom

REFERENCES:
- [Derived] De Doncker W, Ondobaka S, Kuppuswamy A. Effect of transcranial direct current stimulation on post-stroke fatigue. J Neurol. 2021 Aug;268(8):2831-2842. doi: 10.1007/s00415-021-10442-8. Epub 2021 Feb 17. PMID 33598767